CLINICAL TRIAL: NCT01315665
Title: Evaluation of the Effect of Sulforaphane in Broccoli Sprouts on Nrf2 Activation, Measures of Oxidative Stress, and Neutrophil Migration to Mucosal Surfaces in Healthy and CF Subjects
Brief Title: Effect of Sulforaphane in Broccoli Sprouts on Nrf2 Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, James F. Chmiel, Associate Professor of Pediatrics, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UHCMC-CFRC-2011-01
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Cystic Fibrosis
Keywords: broccoli sprouts; sulforaphane; triterpenoid; Nrf2 activation; cystic fibrosis; healthy volunteers; anti-inflammatory
MeSH Terms: conditions — Cystic Fibrosis | interventions — sulforaphane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy volunteers (Experimental): 100 grams of raw broccoli sprouts once daily for 5 consecutive days
  Interventions: Dietary Supplement: Broccoli sprouts
- Subjects with cystic fibrosis (Experimental): 100 grams of raw broccoli sprouts once daily for 5 consecutive days
  Interventions: Dietary Supplement: Broccoli sprouts

INTERVENTIONS:
Dietary Supplement: Broccoli sprouts — Subjects (both healthy volunteers and subjects with cystic fibrosis) will consume 100 gm of raw broccoli sprouts once daily for 5 consecutive days.
  Other Names: sulforaphane

SUMMARY:
The purpose of this study to investigate the effect of sulforaphane from macerated broccoli sprouts in humans and to evaluate less invasive methods of assessing potential anti-inflammatory drugs in CF.

DETAILED DESCRIPTION:
The hypothesis to be tested is that sulforaphane consumed from macerated broccoli sprouts will activate Nrf2, reduce oxidative metabolites and reduce neutrophils in the oral mucosa after 5 days of therapy in healthy volunteers and CF subjects.

The study requires 6 brief outpatient visits over 8 days. Study procedures include medical history, height, weight, vital signs, blood and urine collection, nasal curettage, saline mouthwash, and ingestion of broccoli sprouts (100 gm of 3 to 5 day old raw broccoli sprouts once daily for 5 consecutive days).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers and patients with cystic fibrosis ≥ 18 < 50 years of age
* Healthy volunteers must be in general good health as determined by a medical history
* CF subjects must have a documented diagnosis of CF (positive sweat chloride ≥ 60 mEq/liter, by pilocarpine iontophoresis) and/or a genotype with two identifiable mutations consistent with CF accompanied by one or more clinical features with the CF) phenotype
* CF subjects must have a baseline FEV1 percent predicted > 50% (in the last year, obtained from medical record)
* CF subjects must be clinically stable: free of any acute illness for > 14 days CF subjects must not have been prescribed any new systemic antibiotics for the 14 days prior to enrollment
* Ability to provide written informed consent
* Ability to adhere to the protocol

Exclusion Criteria:

* Use of NSAIDS (e.g., ibuprofen) or corticosteroids including inhaled steroids for the 4 weeks prior to enrollment
* Active gingival disease (active tooth or gum disease)
* History of nephrolithiasis or cholelithiasis
* Allergy to broccoli
* Any chronic condition that compromises the participant as determined by medical history
* Pregnancy
* Inability to tolerate the study procedures
* CF subjects: Infected with B. cepacia

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F. Chmiel, MD, MPH, Principal Investigator — Rainbow Babies and Children's Hospital
Locations (1):
- Rainbow Babies and Children's Hospital, Cleveland, Ohio, United States

REFERENCES:
- [Background] Chmiel JF, Berger M, Konstan MW. The role of inflammation in the pathophysiology of CF lung disease. Clin Rev Allergy Immunol. 2002 Aug;23(1):5-27. doi: 10.1385/CRIAI:23:1:005. PMID 12162106
- [Background] Chen J, Kinter M, Shank S, Cotton C, Kelley TJ, Ziady AG. Dysfunction of Nrf-2 in CF epithelia leads to excess intracellular H2O2 and inflammatory cytokine production. PLoS One. 2008;3(10):e3367. doi: 10.1371/journal.pone.0003367. Epub 2008 Oct 10. PMID 18846238
- [Background] Nichols DP, Ziady AG, Shank SL, Eastman JF, Davis PB. The triterpenoid CDDO limits inflammation in preclinical models of cystic fibrosis lung disease. Am J Physiol Lung Cell Mol Physiol. 2009 Nov;297(5):L828-36. doi: 10.1152/ajplung.00171.2009. Epub 2009 Aug 21. PMID 19700644
- [Background] Verhaeghe C, Remouchamps C, Hennuy B, Vanderplasschen A, Chariot A, Tabruyn SP, Oury C, Bours V. Role of IKK and ERK pathways in intrinsic inflammation of cystic fibrosis airways. Biochem Pharmacol. 2007 Jun 15;73(12):1982-94. doi: 10.1016/j.bcp.2007.03.019. Epub 2007 Mar 24. PMID 17466952
- [Background] Li J, Johnson XD, Iazvovskaia S, Tan A, Lin A, Hershenson MB. Signaling intermediates required for NF-kappa B activation and IL-8 expression in CF bronchial epithelial cells. Am J Physiol Lung Cell Mol Physiol. 2003 Feb;284(2):L307-15. doi: 10.1152/ajplung.00086.2002. Epub 2002 Sep 27. PMID 12388360
- [Background] Escotte S, Tabary O, Dusser D, Majer-Teboul C, Puchelle E, Jacquot J. Fluticasone reduces IL-6 and IL-8 production of cystic fibrosis bronchial epithelial cells via IKK-beta kinase pathway. Eur Respir J. 2003 Apr;21(4):574-81. doi: 10.1183/09031936.03.00031803. PMID 12762338
- [Background] Lands LC, Stanojevic S. Oral non-steroidal anti-inflammatory drug therapy for cystic fibrosis. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD001505. doi: 10.1002/14651858.CD001505.pub2. PMID 17943753
- [Background] Flume PA, O'Sullivan BP, Robinson KA, Goss CH, Mogayzel PJ Jr, Willey-Courand DB, Bujan J, Finder J, Lester M, Quittell L, Rosenblatt R, Vender RL, Hazle L, Sabadosa K, Marshall B; Cystic Fibrosis Foundation, Pulmonary Therapies Committee. Cystic fibrosis pulmonary guidelines: chronic medications for maintenance of lung health. Am J Respir Crit Care Med. 2007 Nov 15;176(10):957-69. doi: 10.1164/rccm.200705-664OC. Epub 2007 Aug 29. PMID 17761616
- [Background] Oermann CM, Sockrider MM, Konstan MW. The use of anti-inflammatory medications in cystic fibrosis: trends and physician attitudes. Chest. 1999 Apr;115(4):1053-8. doi: 10.1378/chest.115.4.1053. PMID 10208207
- [Background] Konstan MW. Ibuprofen therapy for cystic fibrosis lung disease: revisited. Curr Opin Pulm Med. 2008 Nov;14(6):567-73. doi: 10.1097/MCP.0b013e32831311e8. PMID 18812834
- [Background] Shishodia S, Sethi G, Konopleva M, Andreeff M, Aggarwal BB. A synthetic triterpenoid, CDDO-Me, inhibits IkappaBalpha kinase and enhances apoptosis induced by TNF and chemotherapeutic agents through down-regulation of expression of nuclear factor kappaB-regulated gene products in human leukemic cells. Clin Cancer Res. 2006 Mar 15;12(6):1828-38. doi: 10.1158/1078-0432.CCR-05-2044. PMID 16551868
- [Background] Ahmad R, Raina D, Meyer C, Kharbanda S, Kufe D. Triterpenoid CDDO-Me blocks the NF-kappaB pathway by direct inhibition of IKKbeta on Cys-179. J Biol Chem. 2006 Nov 24;281(47):35764-9. doi: 10.1074/jbc.M607160200. Epub 2006 Sep 24. PMID 16998237
- [Background] Dinkova-Kostova AT, Liby KT, Stephenson KK, Holtzclaw WD, Gao X, Suh N, Williams C, Risingsong R, Honda T, Gribble GW, Sporn MB, Talalay P. Extremely potent triterpenoid inducers of the phase 2 response: correlations of protection against oxidant and inflammatory stress. Proc Natl Acad Sci U S A. 2005 Mar 22;102(12):4584-9. doi: 10.1073/pnas.0500815102. Epub 2005 Mar 14. PMID 15767573
- [Background] Liby K, Hock T, Yore MM, Suh N, Place AE, Risingsong R, Williams CR, Royce DB, Honda T, Honda Y, Gribble GW, Hill-Kapturczak N, Agarwal A, Sporn MB. The synthetic triterpenoids, CDDO and CDDO-imidazolide, are potent inducers of heme oxygenase-1 and Nrf2/ARE signaling. Cancer Res. 2005 Jun 1;65(11):4789-98. doi: 10.1158/0008-5472.CAN-04-4539. PMID 15930299
- [Background] Yates MS, Tauchi M, Katsuoka F, Flanders KC, Liby KT, Honda T, Gribble GW, Johnson DA, Johnson JA, Burton NC, Guilarte TR, Yamamoto M, Sporn MB, Kensler TW. Pharmacodynamic characterization of chemopreventive triterpenoids as exceptionally potent inducers of Nrf2-regulated genes. Mol Cancer Ther. 2007 Jan;6(1):154-62. doi: 10.1158/1535-7163.MCT-06-0516. PMID 17237276
- [Background] Konstan MW, Byard PJ, Hoppel CL, Davis PB. Effect of high-dose ibuprofen in patients with cystic fibrosis. N Engl J Med. 1995 Mar 30;332(13):848-54. doi: 10.1056/NEJM199503303321303. PMID 7503838
- [Background] Konstan MW, Schluchter MD, Xue W, Davis PB. Clinical use of Ibuprofen is associated with slower FEV1 decline in children with cystic fibrosis. Am J Respir Crit Care Med. 2007 Dec 1;176(11):1084-9. doi: 10.1164/rccm.200702-181OC. Epub 2007 Sep 13. PMID 17872492
- [Background] Chmiel JF, Konstan MW. Inflammation and anti-inflammatory therapies for cystic fibrosis. Clin Chest Med. 2007 Jun;28(2):331-46. doi: 10.1016/j.ccm.2007.02.002. PMID 17467552
- [Background] Konstan MW, Krenicky JE, Finney MR, Kirchner HL, Hilliard KA, Hilliard JB, Davis PB, Hoppel CL. Effect of ibuprofen on neutrophil migration in vivo in cystic fibrosis and healthy subjects. J Pharmacol Exp Ther. 2003 Sep;306(3):1086-91. doi: 10.1124/jpet.103.052449. Epub 2003 Jun 13. PMID 12807998

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: Healthy volunteers
  Broccoli sprouts: Healthy volunteers will consume 100 gm of raw broccoli sprouts once daily for 5 consecutive days.
- Subjects With Cystic Fibrosis: Subjects with cystic fibrosis
  Broccoli sprouts: Subjects with cystic fibrosis will consume 100 gm of raw broccoli sprouts once daily for 5 consecutive days.
Period: Overall Study
Arm/Group | Healthy Volunteers | Subjects With Cystic Fibrosis
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Subjects With Cystic Fibrosis | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 5 | 15
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 5 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Nrf2 Activation in Nasal Epithelial Cells
Description: Number of subjects with activated Nrf-2 in the cytoplasm of nasal epithelial cells after 5 days of study treatment (consuming broccoli sprouts)
Time Frame: Baseline and of end of 5 day treatment period
Measure: Number; unit: participants
Arm/Group | Healthy Volunteers | Subjects With Cystic Fibrosis
Number analyzed (Participants) | 10 | 5
participants
  Baseline | 0 | 0
  Day 5, End of treatment | 4 | 4

2. Secondary Outcome: Measures of Lipid Peroxidation in Nasal Epithelial Cells
Description: Products of lipid peroxidation will be determined by western blot analysis on nasal epithelial cells obtained by curettage after 5 days of study treatment (consuming broccoli sprouts)
Time Frame: End of 5 day treatment period
Population: Data not collected and will not be analyzed.
Arm/Group | Healthy Volunteers | Subjects With Cystic Fibrosis
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Measures of Glutathione From Blood Lymphocytes
Description: Change in lymphocyte glutathione measurements after 5 days of study treatment (consuming broccoli sprouts).
Time Frame: Baseline and end of 5 day treatment period
Population: Not enough blood could be obtained from one of the healthy volunteers. Therefore, glutathione from blood lymphocytes could not be evaluated from that healthy volunteer. With respect to this outcome measure, only results from 9 healthy volunteers are reported.
Measure: Mean (Standard Deviation); unit: Micro Molar
Arm/Group | Healthy Volunteers | Subjects With Cystic Fibrosis
Number analyzed (Participants) | 9 | 5
Micro Molar | 14.3 (25.9) | 4.7 (48.1)

4. Secondary Outcome: Measures of Oxidative Stress in Urine
Description: Change in urine bromotyrosine (measured by mass spectrometry) will be measured after 5 days of study treatment (consuming broccoli sprouts).
Time Frame: Baseline and end of 5 day treatment period
Measure: Mean (Standard Deviation); unit: ng/mg creatinine (Log10)
Arm/Group | Healthy Volunteers | Subjects With Cystic Fibrosis
Number analyzed (Participants) | 10 | 5
ng/mg creatinine (Log10) | 0.09 (0.23) | 0.01 (0.33)

5. Secondary Outcome: Measure of Neutrophil Migration Into the Gingival Crevices
Description: Change in gingival neutrophils measured after 5 days of study treatment (consuming broccoli sprouts). Patients will perform mouthwashes with normal saline. Neutrophil counts will be performed on fresh samples. Acridine orange will be added to the saline rinses and neutrophils will be counted under the microscope.
Time Frame: Baseline and end of 5 day treatment period
Measure: Mean (Standard Deviation); unit: Neutrophils/mL (Log10)
Arm/Group | Healthy Volunteers | Subjects With Cystic Fibrosis
Number analyzed (Participants) | 10 | 5
Neutrophils/mL (Log10) | -0.06 (0.14) | -0.02 (0.04)

ADVERSE EVENTS:
Arm/Group | Healthy Volunteers | Subjects With Cystic Fibrosis
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 8/10 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers (N=10) | Subjects With Cystic Fibrosis (N=5)
Nausea (Gastrointestinal disorders) | 4 (7) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 3 (6) | 0 (0)
Blood in urine (Renal and urinary disorders) | 0 (0) | 1 (1)
Emesis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gas (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Heartburn (Gastrointestinal disorders) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No